CLINICAL TRIAL: NCT07205393
Title: Phase One Cardiac Rehabilitation Outcomes Post Valve Replacement Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa yussuf abo zaid, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T_INT_11/2024_553
Record Dates: First submitted 2025-09-23; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Valve Replacement Surgery
Keywords: Cardiac rehabilitation; Valve replacement; Spirometry measures
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation (Other): The intervention group underwent the cardiac rehabilitation program from the first day following surgery regarding the clinical guideline for rehabilitation in patients with cardiovascular disease.17 This rehabilitation exercise program formed of breathing exercises, lower and upper extremity exercises in bed, sitting on the edge of the bed, standing at the bedside, and walking around the bed and for 100 m in the ward. The patient performed three sessions per day, with approximately 20 minutes each time. After the rehabilitation exercise, patients continued with gait practice for up to 500 m and carried out endurance training by using a stationary bike in the rehabilitation center of the hospital.
  The sessions continued until they were discharged from the hospital (approximately 5 to 6 days post operative). The intensity of physical activity was limited by clinical conditions and activity tolerance, and monitored and assessed by physical therapists, plus routine clinical care.
  Interventions: Other: Cardiac rehabilitation; Other: Routine clinic care
- Control group (Other): The control group did not joined any rehabilitation program and only received routine clinical care during the duration of the hospital stay (approximately 5 to 6 days post operative).
  Data collection The investigators assessed all patients on the day before surgery (baseline assessment) and the day of hospital discharge.
  Interventions: Other: Routine clinic care

INTERVENTIONS:
Other: Cardiac rehabilitation — The intervention group underwent the cardiac rehabilitation program from the first day following surgery regarding the clinical guideline for rehabilitation in patients with cardiovascular disease.17 This rehabilitation exercise program formed of breathing exercises, lower and upper extremity exercises in bed, sitting on the edge of the bed, standing at the bedside, and walking around the bed and for 100 m in the ward. The patient performed three sessions per day, with approximately 20 minutes each time. After the rehabilitation exercise, patients continued with gait practice for up to 500 m and carried out endurance training by using a stationary bike in the rehabilitation center of the hospital.
  The essions continued until they were discharged from the hospital (approximately 5 to 6 days post operative). The intensity of physical activity was limited by clinical conditions and activity tolerance, and monitored and assessed by physical therapists. Plus routine clinical care
  Arms: Cardiac rehabilitation
Other: Routine clinic care — The control group did not joined any rehabilitation program and only received routine clinical care during the duration of the hospital stay (approximately 5 to 6 days post operative).

SUMMARY:
Cardiac rehabilitation is a crucial component of postoperative recovery for patients who have received valve replacement surgery. Aim: This study aimed to evaluate the effectiveness of phase one cardiac rehabilitation in improving cardiovascular function, pulmonary capacity, functional ability, and quality of life.

DETAILED DESCRIPTION:
A 60 patients aged 40 to 60 years who had received mitral or aortic valve replacement were allocated randomly into two groups equal in numbers, the first one (cardiac rehabilitation group) participated in a phase one cardiac rehabilitation program comprising supervised physical exercises and respiratory training, the second one (control group) underwent routine physical therapy program. The outcomes were oxygen saturation measurements, spirometry measures and Six minutes walk test. All measured variables were evaluated before and after six consecutive weeks of rehabilitation for all patients.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria was elective mitral or aortic valve replacement
* and to be hemodynamically stable to qualify for a structured rehabilitation program.
* Being able to understand and complete measurements.
* And provide informed written consent.

Exclusion Criteria:

* Patient with ischemic heart disease before surgery.
* Those with severe musculoskeletal system disorders.
* Patients who had persistent or paroxysmal atrial fibrillation.
* Individuals with severe heart failure.
* uncontrolled arrhythmias.
* Comorbidity complicating physical activity or other contraindications to phase one cardiac rehabilitation and Patients who underwent an emergency surgical intervention.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation. | 5 to 6 days
  Oxygen saturation: (2700 Branshaj, Denemark).
FVC | 5 to 6 days
  Forced vital capacity (FVC)
FEV1 | 5 to 6 days
  forced expiratory volume in the first second (FEV1)
FEV1/FVC. | 5 to 6 days
  The ratio of FEV1 on FVC.

SECONDARY OUTCOMES:
The 6-Minute Walk Test (6MWT) | 5 to 6 days
  The 6-Minute Walk Test (6MWT): We performed the 6-minute walking test (6MWT), which involved measurement of the 6-minute walking distance and is a submaximal functional test indicative of performing daily activities.18 The safety and feasibility of this test have led to its use in cardiovascular rehabilitation.

CONTACTS AND LOCATIONS:
Locations (1):
- South valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No
I will not share it outside the primary research group.